CLINICAL TRIAL: NCT04787510
Title: COVID-19 Disease and Coagulopathy: Assessment of Clotting Factor Levels in Patients With SARS-CoV-2 Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Collaborators: INTERNAL MEDICINE DEPARTMENT, 1ST WARD (Unknown)
Responsible Party: Principal Investigator, Liontos Angelos, CONSULTANT OF INTERNAL MEDICINE, University Hospital, Ioannina
Other Study IDs: 895/23-12-2020
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: SARS-COV2 Infection; COVID-19 Disease; Hospitalized Patients
MeSH Terms: conditions — COVID-19 | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — PLASMA AND CLOTTING FACTORS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: low molecular weight Heparin as standard of care treatment — STANDARD OF CARE

SUMMARY:
Effect of Covid-19 disease in clotting factors levels in hospitalized patients

DETAILED DESCRIPTION:
Effect of Covid-19 disease in clotting factors levels in hospitalized patients positive for sars-cov2 infection.

Association between clotting factors levels and disease severity,morbidity and mortality in these patients.

Effect of anticoagulant therapy in the clotting factors' levels in these patients

ELIGIBILITY:
Inclusion Criteria:

* AGE> 18
* SINGED INFORMED CONSENT FORM
* POSITIVE PCR TEST FOR SARS-COV2 INFECTION
* FINDINGS IN CXR OR CT OF THE LUNGS CONSISTENT WITH INFECTION OF LOWER RESPIRATORY TRACT

Exclusion Criteria:

* AGE<18
* DENIAL TO PROVIDE INFORMED CONSENT FORM
* HISTORY OF MALIGNANCY
* PRIOR USE OF ANTICOAGULANT THERAPY
* PRIOR USE OF STEROIDS LONGER THAN 14 DAYS
* LACTATION-PREGNANCY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL ELIGIBLE PATIENTS AS DEFINED BY CRITERIA
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
EFFECT OF COVID-19 DISEASE IN CLOTTING FACTORS | 6 MONTHS
  leves of cloting factors before and after treatment with LMWH

CONTACTS AND LOCATIONS:
Overall Officials: HARALAMPOS MILIONIS, PROFESSOR, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University General Hospital of Ioannina, Ioannina, Epirus, Greece